CLINICAL TRIAL: NCT04470232
Title: Transcultural and Psychometric Validation of SUSHI and HOOS-12 Scores in Patients With Coxofemoral Pathologies
Acronym: HIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Lariboisière Hospital (Unknown); Saint-Gregoire Private Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20_RIPH3-03
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2021-12

CONDITIONS: Coxofemoral Pathologies
Keywords: Coxofemoral pathologies; Self assessment questionnaire; Super Simple Hip score (SUSHI-score); Hip disability and Osteoarthritis Outcome Score (HOOS score); Transcultural validation; Psychometric validation; Hip and Groin score (HAGOS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with coxofemoral pathologies: For the transcultural validation, a french version of the 2 self-assessment questionnaires, SUSHI-score and the HOOs-12 score will be produced.
  For the psychometric validation, 120 patients with coxofemoral pathologies will pass the two questionnaires. The HAGOS (Hip and Groin Score) questionnaire will be also passed by the subject, for the convergent validity.
  Interventions: Other: Self-assessment questionnaires

INTERVENTIONS:
Other: Self-assessment questionnaires — 120 patients with coxofemoral pathologies will pass the SUSHI-score and the HOOS-12 score questionnaires.
  The HAGOS (Hip and Groin Score) questionnaire will be also passed by the subject, for the convergent validity.

SUMMARY:
The management of coxofemoral pathologies is constantly increasing.

In addition to degenerative hip pathology, the orthopedic surgeon is now confronted with pathologies such as femoro-acetabular conflict, pathologies of the gluteus medius and pathologies of the labrum whose early management limits arthritis degeneration. These pathologies are mainly encountered in young subjects (<60 years).

Self-questionnaires play an important role in understanding patients' point of view on the impact of their coxofemoral pathologies and also allow an assessment of their condition after treatment.

For the evaluation of coxofemoral pathologies in the young subject (<60 years) the Super Simple Hip score (SUSHI-score) was developed and validated.

In the elderly subject with hip osteoarthritis, the HOOS score has the advantage of specifically measuring pain, symptoms, function and quality of life, but is made up of 40 items and is often considered rather heavy to submit. However, it has recently been simplified and the HOOS-12 (HOOS score with 12 items) has been developed and validated.

These two scores are useful in current clinical practice but they are only validated in English.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age greater than or equal to 18 years old),
* Patient with coxofemoral pathology,
* Patient having been informed of the research,
* Patient agreeing to participate in the study.

Exclusion Criteria:

* Minor patient,
* Pregnant woman,
* Patient out of state to agree to participate in the study,
* Patient unable to answer a self-assessment questionnaire,
* Patient under justice, guardianship or curatorship,
* Patient who refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a coxofemoral pathology.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Transcultural validation of the SUSHI-score and HOOS-12 score questionnaire | 1 month
  It will be a question of obtaining a version translated into French. The translated version tested on a small group of patients (15) will be submitted to the author of the original version of the tool, along with a report highlighting and explaining all the modifications and difficulties noted by a group of experts.
Psychometric validation of the SUSHI-score and HOOS-12 score questionnaire | 12 months
  Questionnaires will be passed by 120 subjects. Following parameters will be measured: feasibility and acceptability, validity, reliability, and sensitivity to change.

CONTACTS AND LOCATIONS:
Locations (3):
- France (2):
  - Hôpital Lariboisière - AP-HP, Paris
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
- CHU of Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No